CLINICAL TRIAL: NCT01754207
Title: Evaluation of the 755nm Alexandrite Laser for the Treatment of Tattoos
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cynosure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYN11-PICO-D-A-TAT
Record Dates: First submitted 2012-12-18; First posted 2012-12-21 (Estimated); Results first posted 2020-12-16 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-11

CONDITIONS: Tattoos
MeSH Terms: interventions — Lasers, Solid-State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 755nm Alexandrite Laser (Experimental): 755nm Alexandrite Laser
  Interventions: Device: 755nm Alexandrite Laser; Device: 755nm Alexandrite Laser with CAP Array

INTERVENTIONS:
Device: 755nm Alexandrite Laser — 755nm Alexandrite Laser
Device: 755nm Alexandrite Laser with CAP Array — 755nm Alexandrite Laser with CAP Array

SUMMARY:
The purpose of this study is to collect further data on the safety and efficacy of removing unwanted non cosmetic tattoos (including recalcitrant) using the 755nm Alexandrite laser.

ELIGIBILITY:
Inclusion Criteria:

1. Is a healthy male or female between 18 and 85 years old.
2. Has unwanted non-cosmetic tattoo(s) and wishes to undergo laser treatments to remove them.
3. Is willing to consent to participate in the study.
4. Is willing to comply with all requirements of the study including being photographed, following post treatment care and attending all treatment and follow up visits

Exclusion Criteria:

1. Is hypersensitive to light exposure.
2. Has active localized or systemic infection.
3. Is taking medication(s) for which sunlight is a contraindication.
4. Has a history of squamous cell carcinoma or melanoma.
5. Has a history of keloid scarring.
6. Has used oral isotretinoin (Accutane®) within 12 months of initial treatment or plans on using during the course of the study. Note: Skin must regain its normal degree of moisture prior to treatment.
7. Has a history of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or use of immunosuppressive medications.
8. Is female and pregnant, has been pregnant within the last 3 months, is currently breast feeding or planning a pregnancy during the study period.
9. Is allergic to lidocaine, tetracaine or Xylocaine with epinephrine.
10. Has any other reason determined by the physician to be ineligible to participate in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-12; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Krantz, Study Director — Cynosure, Inc.
Locations (1):
- Skin Care Physicians, Chestnut Hill, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 755nm Alexandrite Laser
Started | 20
Completed | 17
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | 755nm Alexandrite Laser
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Caucasian | 18
  Race/Ethnicity: Hispanic | 1
  Race/Ethnicity: African American | 1
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — The Fitzpatrick Skin Score is used to determine skin color. It is a numerical system that classifies skin into six types (Type I, Type II, Type III, Type IV, Type V and Type VI) based on the numerical score achieved (ranging from 0 to 36). The lower the score (and skin type number), the fairer the skin. The higher the score (and skin type number), the more deeply pigmented the skin is.
  The scale comes from this source:
  Gupta, Sharma. Skin typing: Fitzpatrick grading and others. Clinics in Dermatology. 2019;37(5):430-436. doi:10.1016/j.clindermatol.2019.07.010
  Participants
    Fitzpatrick Skin Score I | 4
    Fitzpatrick Skin Score II | 9
    Fitzpatrick Skin Score III | 6
    Fitzpatrick Skin Score IV | 1
    Fitzpatrick Skin Score V | 0
    Fitzpatrick Skin Score VI | 0

OUTCOME MEASURES:

1. Primary Outcome: Tattoo Clearance Using Photographic Evaluation
Description: 2D photography comparing pre and post treatment photos, where the percentage of tattoo clearance between the photos was determined by the evaluator.
Time Frame: up to 3 months post last treatment
Measure: Count of Units; unit: Tattoos
Units Other Than Participants: Tattoos
Arm/Group | 755nm Alexandrite Laser
Number analyzed (Participants) | 17
Number analyzed (Tattoos) | 23
Tattoos
  >75% clearance | 15
  51-74% clearance | 6
  <25% clearance | 2

ADVERSE EVENTS:
Time Frame: Adverse Events occurring were captured for the study duration, around 12 months.
Description: Adverse Events listed under "other" were monitored/assessed without regard to the specific Adverse Event Term.
Arm/Group | 755nm Alexandrite Laser
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 20/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 755nm Alexandrite Laser (N=20)
Pain (Nervous system disorders) | 9
Erythema (Skin and subcutaneous tissue disorders) | 16
Pinpoint Bleeding (Skin and subcutaneous tissue disorders) | 10
Edema (Skin and subcutaneous tissue disorders) | 16
Crusting (Skin and subcutaneous tissue disorders) | 15
Scabbing (Skin and subcutaneous tissue disorders) | 14
Blistering (Skin and subcutaneous tissue disorders) | 16
Purpura (Skin and subcutaneous tissue disorders) | 6
Hypopigmentation (Skin and subcutaneous tissue disorders) | 2
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 3
Bruising (Skin and subcutaneous tissue disorders) | 1
Other (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI cannot disclose confidential or proprietary information until after it becomes generally known or available to the public.